CLINICAL TRIAL: NCT06990815
Title: The Immediate Effect of Kinesio Taping on Pain, Menstrual Symptoms, Fear of Movement, and Sleep Quality in Primary Dysmenorrhea: A Randomized Sham-Controlled Trial
Brief Title: Immediate Effects of Kinesio Taping in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Assos. Prof, Okan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12.4.2023/6
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Primary Dysmenorrhea
Keywords: Kinesio Taping; Pain; Menstrual Symptoms; Fear of Movement; Sleep Quality
MeSH Terms: conditions — Pain; Kinesiophobia; Sleep Initiation and Maintenance Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Group (Experimental)
  Interventions: Other: Kinesio Taping
- Sham Control Group (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: Kinesio Taping — In the application over the sacrum, one I-strip of kinesio tape will be applied with 25% tension using the fascia correction technique, which requires oscillatory movements between the tape and the skin.
  In the application over the suprapubic region, two I-strips will be applied with 25% tension, also using the fascia correction technique, involving oscillations between the tape and the skin.
  Arms: Kinesio Taping Group
Other: Sham — In the application over the sacrum, one I-strip will be applied without tension.
  In the application over the suprapubic region, two I-strips will be placed without tension.
  Arms: Sham Control Group

SUMMARY:
Primary dysmenorrhea is characterized by recurrent, cramping lower abdominal pain during menstruation and affects approximately 50% to 90% of women. The etiology of primary dysmenorrhea involves the increased release of prostaglandins and other inflammatory mediators, which cause uterine contractions and reduced blood flow. In addition to pharmacological approaches, non-pharmacological methods also play an important role in the treatment of dysmenorrhea.

Kinesio taping helps relieve pain by reducing pressure on the muscle and supports treatment through various application techniques. It improves local circulation, reduces muscle tension, and alleviates symptoms of primary dysmenorrhea.

The aim of this study is to investigate the effects of kinesio taping on pain, menstrual symptoms, fear of movement, and sleep quality in women with primary dysmenorrhea, and to compare the outcomes with those of a sham taping group.

The hypothesis is that kinesio taping will be more effective than sham taping in improving these parameters in women with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Being a nulliparous woman aged between 18 and 24 years
* Having a diagnosis of primary dysmenorrhea confirmed by a physician,
* Being literate
* Cooperating in completing the assessment scales
* Scoring one or above on the Weissman Scale
* Agreeing to participate in the study
* Having regular menstruation in the last 6 months
* Being willing and voluntary to participate in the research.

Exclusion Criteria:

* Having a diagnosis of secondary dysmenorrhea
* Using contraceptive pills
* Having a history of childbirth or pregnancy
* Having irregular menstrual cycles (menstrual cycle length less than 21 days or longer than 35 days)
* Having any pelvic pathology or history of pelvic surgery
* Having gastrointestinal, urogynecological, autoimmune, psychiatric, neurological diseases, or other chronic pain syndromes.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Being a nulliparous woman aged between 18 and 24 years
Enrollment: 24 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 weeks
  Pain will be assessed using the Visual Analog Scale. On the Visual Analog Scale, a score of '0' indicates no pain, while '10' represents the most unbearable pain on a 10 cm horizontal line. It is a simple, practical, valid, reliable, and reproducible measurement tool.
Menstrual Symptom Questionnaire | 2 weeks
  The Menstrual Symptom Questionnaire (MSQ) was originally developed by Chesney and Tasto in 1975 to evaluate menstrual pain and related symptoms. Participants rate the severity of symptoms they experience during menstruation on a scale from 1 (never) to 5 (always).
  In this scale:
  Items 1-13 assess negative effects, Items 14-19 assess menstrual pain symptoms, and Items 20-22 assess coping methods. As the average score of each subscale increases, it indicates a higher severity of menstrual symptoms related to that subscale.
Menstrual Attitude and Behavior Scale | 2 weeks
  The Menstrual Attitude and Behavior Scale will be used to assess individuals' attitudes and behaviors during the menstrual period. This scale, also known as the Menstrual Attitude Questionnaire, consists of 33 items divided into five subscales:
  Menstruation as a debilitating event - 12 items Menstruation as a bothersome event - 6 items Menstruation as a natural event - 5 items Anticipation of the onset of menstruation - 5 items Denial of menstrual effects - 7 items Each subscale provides insight into specific attitudes and perceptions related to menstruation.
Tampa Scale of Kinesiophobia | 2 weeks
  Fear of movement will be assessed using the Tampa Scale of Kinesiophobia. The scale uses a 4-point Likert-type scoring system, and the total score ranges from 17 to 68.
  Higher scores indicate a greater fear of movement.
Richard Campbell Sleep Questionnaire | 2 weeks
  The Richard Campbell Sleep Questionnaire was developed by Richards in 1987 to assess sleep depth, time taken to fall asleep, number of awakenings, duration of wakefulness after sleep onset, sleep quality, and environmental noise level.
  It consists of 6 items, each evaluated using a visual analog scale ranging from 0 to 100. A score between 0-25 indicates very poor sleep, while a score between 76-100 reflects very good sleep. The total score is calculated based on 5 items; the 6th item, which evaluates environmental noise level, is excluded from the total score. Higher total scores indicate better sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided